CLINICAL TRIAL: NCT07350473
Title: Vibration-Assisted Physical Activity for Glycaemic Control in Type-2 Diabetes: A Randomised Controlled Trial in the Kingdom of Saudi Arabia
Brief Title: Effects of Vibration-Assisted Physical Activity in Type-2 Diabetes
Acronym: VIBRANT-KSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Collaborators: University of Jazan (Other Government); University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vibration-Assisted Physical Ac
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Localized Vibration (Experimental)
  Interventions: Device: Localized vibration
- Placebo vibration (Sham Comparator)
  Interventions: Other: Placebo vibration
- Usual care (Other)
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Localized vibration — Participants allocated to the localized vibration group will complete home based sessions five times per week for 12 weeks. Each session will last approximately 60 minutes and will consist of four 10 minute bouts of focal muscle vibration separated by 5 minute seated rest periods. Participants will be seated with hips and knees at roughly 90 degrees and will perform repeated calf raises, executing plantarflexion within an approximate 0-45° range at a cadence of 60 repetitions per minute.
  Arms: Localized Vibration
Other: Placebo vibration — Participants allocated to the placebo group will follow an identical protocol to the active vibration arm, including the same session frequency, activity and durations. However, they will use a sham version of the wearable device that emits only negligible vibration, providing minimal cutaneous sensation without delivering a meaningful therapeutic dose.
  Arms: Placebo vibration
Other: Usual care — Usual care.
  Arms: Usual care

SUMMARY:
The World Health Organization ranks Saudi Arabia as having the 7th highest rate of type-2 diabetes in the world. This therefore makes diabetes the most challenging health problem facing Saudi Arabia. Importantly, physical activity has been shown to improve disease symptoms and overall health in patients with type-2 diabetes. However, findings relating to the prevalence of physical inactivity in the Saudi population confirm that a sedentary lifestyle is on the rise, within physical inactivity levels in adults being 80.5%. Therefore, interventions aimed at reducing physical inactivity using bespoke modalities pertinent to Saudi Arabia are clearly warranted.

There have been no fully powered, placebo-controlled trials of localised wearable calf vibration in T2DM within the Kingdom of Saudi Arabia. The proposed study will address this gap by evaluating a 12 week, home based, seated calf vibration intervention in Saudi adults with T2DM, recruited from the Jazan Diabetes and Endocrinology Center. A three-arm design will compare active localised vibration, a sham vibration condition and usual care.

ELIGIBILITY:
Inclusion Criteria:

* Clinically established diagnosis of type-2 diabetes for at least 12 months
* Previously sedentary
* Knowledgeable about hypoglycaemia
* Aged over 18 years
* Capacity to give informed consent.

Exclusion Criteria:

* Cognitive impairment precluding consent or participation
* Pregnancy
* Additional medical conditions that prevent safe physical activity (e.g. severe arthritis or advanced heart failure)
* Enrolment in any other clinical trial designed to influence type-2 diabetes symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
HBA1c (Glycated hemoglobin) | Baseline
  Glycated hemoglobin is a form of hemoglobin that is chemically linked to a sugar. This parameter will be obtained via a venous blood sample.
HBA1c (Glycated hemoglobin) | 12 weeks
  Glycated hemoglobin is a form of hemoglobin that is chemically linked to a sugar. This parameter will be obtained via a venous blood sample.
HBA1c (Glycated hemoglobin) | 24 weeks
  Glycated hemoglobin is a form of hemoglobin that is chemically linked to a sugar. This parameter will be obtained via a venous blood sample.

SECONDARY OUTCOMES:
WHO Well-Being Index (WHO-5) | Baseline
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. A score of 0 represents the worst imaginable well-being and 100 represents the best imaginable well-being.
WHO Well-Being Index (WHO-5) | 12 weeks
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. A score of 0 represents the worst imaginable well-being and 100 represents the best imaginable well-being.
WHO Well-Being Index (WHO-5) | 24 weeks
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. A score of 0 represents the worst imaginable well-being and 100 represents the best imaginable well-being.
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  The Patient Health Questionnaire-9 (PHQ-9) is the depression module, which has nine questions ranging from "0" (not at all) to "3" (nearly every day). The scoring is interpreted as 0-4 no depression symptoms, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depression symptoms.
Patient Health Questionnaire-9 (PHQ-9) | 12 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is the depression module, which has nine questions ranging from "0" (not at all) to "3" (nearly every day). The scoring is interpreted as 0-4 no depression symptoms, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depression symptoms.
Patient Health Questionnaire-9 (PHQ-9) | 24 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is the depression module, which has nine questions ranging from "0" (not at all) to "3" (nearly every day). The scoring is interpreted as 0-4 no depression symptoms, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depression symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | 24 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Physical fitness | Baseline
  Physical fitness will be examined via the Chester Step test.
Physical fitness | 12 weeks
  Physical fitness will be examined via the Chester Step test.
Physical fitness | 24 weeks
  Physical fitness will be examined via the Chester Step test.
Fasting glucose | Baseline
  Fasting glucose levels will be examined via a venous blood sample.
Fasting glucose | 12 weeks
  Fasting glucose levels will be examined via a venous blood sample.
Fasting glucose | 24 weeks
  Fasting glucose levels will be examined via a venous blood sample.
Systolic blood pressure | Baseline
  Systolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Systolic blood pressure | 12 weeks
  Systolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Systolic blood pressure | 24 weeks
  Systolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Diastolic blood pressure | Baseline
  Diastolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Diastolic blood pressure | 12 weeks
  Diastolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Diastolic blood pressure | 24 weeks
  Diastolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Body mass | Baseline
  Body mass in kg measured via an electric scale.
Body mass | 12 weeks
  Body mass in kg measured via an electric scale.
Body mass | 24 weeks
  Body mass in kg measured via an electric scale.
Body mass index | Baseline
  Body mass index will be quantified using the standard body mass index equation using measures of body mass and stature.
Body mass index | 12 weeks
  Body mass index will be quantified using the standard body mass index equation using measures of body mass and stature.
Body mass index | 24 weeks
  Body mass index will be quantified using the standard body mass index equation using measures of body mass and stature.
Triglyceride-glucose index | Baseline
  The triglyceride-glucose index will be calculated using a logarithm of the fasting triglyceride and glucose indices.
Triglyceride-glucose index | 12 weeks
  The triglyceride-glucose index will be calculated using a logarithm of the fasting triglyceride and glucose indices.
Triglyceride-glucose index | 24 weeks
  The triglyceride-glucose index will be calculated using a logarithm of the fasting triglyceride and glucose indices.
Total cholesterol | Baseline
  This parameter will be obtained via a venous blood sample.
Total cholesterol | 12 weeks
  This parameter will be obtained via a venous blood sample.
Total cholesterol | 24 weeks
  This parameter will be obtained via a venous blood sample.
HDL cholesterol | Baseline
  This parameter will be obtained via a venous blood sample.
HDL cholesterol | 12 weeks
  This parameter will be obtained via a venous blood sample.
HDL cholesterol | 24 weeks
  This parameter will be obtained via a venous blood sample.
LDL cholesterol | Baseline
  This parameter will be obtained via a venous blood sample.
LDL cholesterol | 12 weeks
  This parameter will be obtained via a venous blood sample.
LDL cholesterol | 24 weeks
  This parameter will be obtained via a venous blood sample.
Triglycerides | Baseline
  This parameter will be obtained via a venous blood sample.
Triglycerides | 12 weeks
  This parameter will be obtained via a venous blood sample.
Triglycerides | 24 weeks
  This parameter will be obtained via a venous blood sample.

IPD SHARING:
Plan to Share IPD: No